CLINICAL TRIAL: NCT05183945
Title: Preoperative Computed Tomography-guided Localization for Lung Nodules: Localization Needle Versus Coil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xuzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20211221005
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Lung; Node
Keywords: Lung nodule; Localization; Coil; Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Localization needle insertion (Experimental): Patients undergo localization needle insertion on day 1.
  Interventions: Device: Localization needle
- Coil insertion (Active Comparator): Patients undergo coil insertion on day 1.
  Interventions: Device: Coil

INTERVENTIONS:
Device: Localization needle — A localization needle which is used for preoperative localization of lung nodules.
  Arms: Localization needle insertion
Device: Coil — A coil which is used for preoperative localization of lung nodules.
  Arms: Coil insertion

SUMMARY:
Preoperative computed tomography-guided localization can improve technical success rates associated with sublobar lung nodule resection conducted via video-assisted thoracoscopic surgery. This study sought to compare the clinical efficacy of computed tomography-guided localization needle and coil insertion as approaches to preoperative lung nodule localization.

DETAILED DESCRIPTION:
Lung nodules are frequently diagnosed and often exhibit a high potential for malignancy such that they are commonly diagnosed and treated via video-assisted thoracic surgery approaches. Preoperative computed tomography-guided localization strategies are commonly employed to improve the successful rate of video-assisted thoracic surgery-guided sublobar (wedge or segmental) resection procedures. One recent meta-analysis found coil localization to be associated with the lowest rate of complications of tested localization materials. Hook-wire has also been widely used due to its simple placement approaches. However, a number of recent reports have suggested that hook-wire insertion approaches are associated with an increased potential for frequent and potentially severe complications.

The use of a novel lung nodule localization needle strategy based on the modification of this previously described hook-wire approach has recently been employed in clinical contexts. Such localization needles have the potential to incur lower rates of detachment and complications relative to the hook-wire strategy without resulting in an increase in localization difficulty. The relative clinical efficacy of localization needle-based strategies compared to that of other localization materials, however, has yet to be established in the context of lung nodule localization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with lung nodules;
2. Patients with an intermediate-to-high risk of malignancy as established based upon radiological and clinical findings.

Exclusion Criteria:

1. Lung nodule < 5 mm;
2. Calcification nodules;
3. Lung nodule which decreased in size at time of follow-up;
4. Patients with distant metastases or other severe comorbidities.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Technical success of localization | From the date of randomization until the date of first documented failure localization from any cause, assessed up to 7 day.
  Lung nodule localization is considered technically successful if the coil tail or marked line can be visible during the video-assisted thoracoscopic surgery. procedure

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Chi Li, MD, Principal Investigator — Xuzhou Central Hospital
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.

REFERENCES:
- [Background] Fu YF, Zhang M, Wu WB, Wang T. Coil Localization-Guided Video-Assisted Thoracoscopic Surgery for Lung Nodules. J Laparoendosc Adv Surg Tech A. 2018 Mar;28(3):292-297. doi: 10.1089/lap.2017.0484. Epub 2017 Nov 14. PMID 29135327